CLINICAL TRIAL: NCT04038411
Title: Single-arm, Multi-center Clinical Study of PD-1 Antibody, Chidamide, Lenalidomide and Etoposide for Relapsed or Refractory Natural Killer/T Cell Lymphoma
Brief Title: PD-1 Antibody, Chidamide, Lenalidomide and Etoposide for Relapsed or Refractory NK/T Cell Lymphoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mingzhi Zhang (Other)
Responsible Party: Sponsor-Investigator, Mingzhi Zhang, the director of oncology department of the first affiliated hospital, Zhengzhou University
Organization: Zhengzhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hnslblzlzx2019070202
Record Dates: First submitted 2019-07-02; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-04

CONDITIONS: NK/T Cell Lymphoma
Keywords: PD-1 Antibody; chidamide; lenalidomide; etoposide; NK/T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Lenalidomide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 Antibody, chidamide, lenalidomide and etoposide (Experimental): PD-1 Antibody: 240mg, d1, Chidamide: 20mg, twice a week, Lenalidomide: 25mg, d1-14 Etoposide:100mg/m2, d1-3 and 21 days made one treatment cycle.
  Interventions: Drug: PD-1 Antibody, chidamide, lenalidomide and etoposide

INTERVENTIONS:
Drug: PD-1 Antibody, chidamide, lenalidomide and etoposide — PD-1 blocking antibody inhibits PD-1. Chidamide is an histone deacetylase inhibitor. Lenalidomide is a potent inhibitor of TNF-α. Etoposide inhibits DNA synthesis by forming a complex with topoisomerase II and DNA.

SUMMARY:
To observe the safety, tolerability and clinical effects of PD-1 Antibody, Chidamide, Lenalidomide and Etoposide in Relapsed or Refractory NK/T cell Lymphoma.

DETAILED DESCRIPTION:
This is a prospective, open-label, one-arm, multicenter clinical trial, aimed to evaluate the safety, tolerability, and efficacy of PD-1 Antibody, Chidamide, Lenalidomide and Etoposide in Relapsed or Refractory NK/T cell Lymphoma. A total of 50 patients are planned to be enrolled into the study. The primary end points are objective responder rate (ORR) and progression free survival(PFS) and the secondary end points include overall survival(OS) , and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. age:14-65 years;Eastern Cooperative Oncology Group (ECOG)score≤2;expected survival≥3 months;
2. patients with NK/T Cell Lymphoma diagnosed by immuno-histochemistry (IHC) or fluorescence in situ hybridization (FISH);
3. Refractory or relapse after at least 2 regimen;
4. Once the patient received radiotherapy, need to be more than 3 months away from this treatment, and it is a non-primary recurrence;
5. No chemotherapy contraindications: hemoglobin ≥ 100g / L, absolute neutrophil count ≥ 1.5 × 109 / L, platelets ≥ 80 × 109 / L, ALT, AST ≤ 2 times the upper limit of normal, serum total bilirubin ≤ 1.5 times normal Upper limit, serum creatinine ≥ 1.5 times normal upper limit, serum protein ≥ 30g / L;
6. At least one measurable lesion;
7. There are no other serious diseases that conflict with this program, and the cardiopulmonary function is normal;
8. Women of childbearing age must have a negative urine or blood pregnancy test, and male patients should be contraceptive during medication;
9. There is no other antitumor treatment, but bisphosphonate for anti-bone metastasis treatment and other symptomatic treatment can be applied;
10. Can understand the situation of this study and sign the informed consent voluntarily

Exclusion Criteria:

1. rejecting providing blood preparation;
2. allergic to drug in this study or with hemophagocytic syndrome;
3. rejecting adopting reliable contraceptive method in pregnancy or lactation period;
4. uncontrolled internal medicine disease(including uncontrolled diabetes,severe incompetence cardiac,lung,liver and pancreas）；
5. with severe infection;
6. with primary or secondary central nervous system tumor invasion;
7. with Chemotherapy or radiotherapy contraindication;
8. ever suffered with malignant tumor;
9. Human immunodeficiency virus (HIV)-positive patients
10. Drug abuse or long-term alcohol abuse that affects the evaluation of test results;
11. Have peripheral nervous system disorder or mental disorder;
12. Patients with immune system diseases;
13. Those who have no legal capacity or whose research is affected by medical or ethical reasons;

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | From date of randomization until the date of first date tumor volume has reduced, assessed up to 36 months
  The proportion of patients whose tumor volume has reduced to a predetermined value and can maintain the minimum time limit is the sum of complete and partial mitigation.

SECONDARY OUTCOMES:
Progression-free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  The time between the start of randomization and the progression of the tumor (any aspect) or (for any reason) death
Overall Survival | From date of randomization until date of death from any cause, assessed up to 36 months
  Time from randomization to death for any reason.

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Department of The First Affilliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No